CLINICAL TRIAL: NCT00225667
Title: Irbesartan for the Prevention of Atrial Arrhythmias and Cardiac Electrical Remodeling in Patients With Hypertension, Permanent Pacemakers and Risk Factors for Developing Atrial Fibrillation
Brief Title: Irbesartan for the Prevention of Atrial Arrhythmias and Cardiac Electrical Remodeling in Patients With Hypertension and Permanent Pacemakers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Connolly, Stuart, M.D. (Individual)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 099104; CTA-099104
Record Dates: First submitted 2005-09-12; First posted 2005-09-26 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-11

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: Atrial Fibrillation; Arrhythmia; Pacemaker, Artificial; Atrial High Rate Episodes; Electrophysiology; Renin-Angiotensin System; Hypertension; Cardiac Remodeling
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Arrhythmias, Cardiac | interventions — Irbesartan

INTERVENTIONS:
Drug: Irbesartan

SUMMARY:
The purpose of this study is to determine whether irbesartan will reduce the rate of recurrent atrial high rate episodes and the development of clinical sustained atrial fibrillation in patients with hypertension and permanent pacemaker.

DETAILED DESCRIPTION:
Patients with permanent pacemakers have a high risk of atrial fibrillation (AF), particularly those with hypertension, sinus node dysfunction, and those with short episodes of atrial arrhythmias, known as atrial high-rate episodes (AHRE). AHRE are felt to be a precursor to AF, and may be both the result and a cause of changs in the atrial electrophysiology, and structure (known as cardiac remodeling)that are associated with the development of AF.

Evaluating this process in human AF has been limited by the cumbersome nature of performing serial, invasive electrophysiologic studies. However, modern pacemakers now permit rapid, non-invasive electrophysiologic testing and can also accurately document AHRE, which allows the convenient study of therapy aimed at preventing the progression from AHRE to overt AF. In addition, this group of patients also affords the ability to evaluate the recurrence of AHRE on the progression of structural and electrical remodeling.

Comparison: Irbesartan compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Sinus Node Dysfunction (with or without AV conduction disturbance)
* Permanent, atrial or dual-chamber pacemaker implanted > 2 months before enrollment and with ability to record and store atrial high-rate episodes, frequency of mode switches and to perform non-invasive electrophysiologic testing
* History of at least 6 AHRE in the last 6 months (rate > 220/min, duration of > 2 minutes
* History of prior diagnosis of hypertension and/or treated for hypertension OR two documented BP > 130/85 (measurements done at least one week apart)

Exclusion Criteria:

* Permanent or persistent AF or more than 6 episodes of symptomatic paroxysmal AF in the previous 6 months
* Documented Cr >200 umol/L and K+ >5.2 mmol/L in the previous 3 months
* Current treatment with a potassium sparing diuretic, unless serum potassium known to be in the normal range
* LV ejection fraction known to be < 40 %
* Moderate or severe mitral regurgitation (3+, 4 +)
* Mitral stenosis of more than mild severity
* Aortic stenosis with mean gradient of > 25 mmHg
* Angina at rest in the last 2 months, or current CCS Class 3 or 4 angina
* Unipolar atrial lead
* Previous AV node ablation
* P-wave amplitude less than 1.5 mV
* Current therapy with an ACE inhibitor, ARB or aldosterone antagonist
* Current or planned (within 6 months) with an anti-arrhythmic medication (amiodarone, sotalol, flecainide, propafenone, quinidine, dofetilide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-12; Study Completion 2007-07

PRIMARY OUTCOMES:
Time to recurrent AHRE ( 220/min for > 2 minutes)

SECONDARY OUTCOMES:
- Frequency of AHRE's (> 220/min for > 2 minutes) Evaluated at randomization, month 1 and 6.
- Development of sustained AF (>30 minutes), documented
by ECG, holter, rhythm strip or pacemaker electrograms
- Electrical Remodeling (AERP,SNRT,paced/sensed p-wave
duration). Evaluated at randomization, months 1 and 6.
- Markers of Inflammation (Plasma CRP,TNF-alpha, D-Dimer,
IL-6, Pro-collagen-III products, BNP,MPO,hsP). Blood collection at randomization and month 6.
- Structural Remodeling (left atrial volume, left
ventricular mass, left ventricular diastolic function. Evaluated at randomization and month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J. Connolly, MD, Principal Investigator — McMaster University; Jeffrey S Healey, MD, Principal Investigator — McMaster University; Carlos A Morillo, MD, Principal Investigator — McMaster University; Stefan H Hohnloser, MD, Principal Investigator — J.W. Goethe University, Frankfurt Germany; Carsten W Israel, MD, Principal Investigator — J.W. Goethe University, Frankfurt Germany
Locations (1):
- Population Health Research Institute of McMaster University, Hamilton, Ontario, Canada